CLINICAL TRIAL: NCT00179881
Title: Thalomid and Carboplatin for the Treatment of Pediatric Brain Stem Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Stewart Goldman, Division Head, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS 1099
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Brain Stem Neoplasms, Primary; Neoplasms, Brain Stem
Keywords: Brain stem glioma
MeSH Terms: conditions — Brain Stem Neoplasms | interventions — Carboplatin; Thalidomide

INTERVENTIONS:
Drug: Carboplatin
Drug: Thalomid
Procedure: External Beam Radiation Therapy

SUMMARY:
Treatment on this study combines two drugs: Thalomid™ (thalidomide) and carboplatin. Thalidomide has been available for many years and has been used to treat many different illnesses. Carboplatin is an effective medicine in killing cancer cells. Thalidomide works by blocking angiogenesis (the process of new blood vessel formation). If a tumor does not have blood vessels providing oxygen and nutrients, it will not be able to grow. This research will look at how combining the effects of thalidomide (preventing tumor growth) with the tumor killing effect of carboplatin effects the long-term outlook for patients with these tumors.

This study will try to find out how well Thalomid™ and carboplatin combined with radiation therapy works in treating children newly diagnosed with brain stem glioma. This study will look at how well Thalomid ™ and carboplatin work in patients with recurrent brain stem glioma. This study will also look at any side effects of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >/= 3 and </= 21 years of age.
* Patients must have a newly diagnosed or progressive brain stem tumor.
* If biopsy has been performed, patients with both high and low grade astrocytomas are eligible.
* Non-histologically confirmed brain stem tumors are eligible. Neuroradiographic confirmation of brain stem glioma is mandatory for study entry.
* Cervicomedullary junction tumors are ineligible.
* Patients with a diagnosis of NF-1 are ineligible.
* Patients must be registered within 6 weeks from diagnosis or recurrence.
* Patients must have life expectancy > 6 weeks.
* Patients must have adequate hematologic and renal function: ANC >1,000/ul, platelets>100,000/ul and creatinine normal for age: </= 0.7 mg/dl (age 3-10yrs.), </= 1.0 mg/dl (11-12yrs.). and </= 1.2 (13-21yrs.).
* Written informed consent must be obtained according to institutional guidelines.
* Pregnant or nursing women are ineligible.
* Patients must be registered within 3 days prior to the start of protocol treatment. Patients must not start treatment until informed consent is given and the patient is registered. Willingness and ability to comply with the FDA-mandated S.T.E.P.S.® program.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Estimated)
Dates: Start 1999-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To determine overall and event free survival for newly diagnosed brain stem glioma with the protocol regimen.
To determine the overall survival and progression free survival of patients with recurrent brain stem glioma.
To determine the toxicity of this drug regimen.

SECONDARY OUTCOMES:
To determine whether the multi-agent chemotherapy regimen of thalidomide and carboplatin, in patients with recurrent brain stem gliomas will extend their survival as compared to historical controls.
To formulate experimentally derived hypothesis in order to establish a basis for future investigational studies.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (6):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospitals and Clinics, Minneapolis, Minnesota
  - Children's Hospitals and Clinics, Saint Paul, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Children's Medical Center, Dayton, Ohio